CLINICAL TRIAL: NCT04218383
Title: Effect of Transcranial Direct Current Stimulation (tDCS) Applied Over the Orbitofrontal Cortex on Impulsivity and Decision Making in Obese Subjects
Brief Title: Transcranial Direct Current Stimulation for Impulsivity and Food-related Impulsivity in Obesity
Acronym: tDCS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Coronavirus pandemic
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REB19-0171
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental: Active Left OFC Group (Active Comparator): 2mA will be applied for 20 minutes with the tDCS anode applied to the left OFC and Cathode applied to the right primary motor cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Comparator: Sham left OFC Group (Sham Comparator): Current will be ramped up for 30s followed by a 30s ramp down to mimic the physical sensation of stimulation and habituation. The anode placed over the left OFC and cathode placed over the right primary motor cortex.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anode placed over the OFC and cathode placed over the right primary motor cortex.
  Other Names: tDCS

SUMMARY:
In this study the investigators aim to assess whether transcranial direct current stimulation (tDCS; a safe non-invasive method for modulating the activity of specific brain regions) when applied over the orbitofrontal cortex (OFC) is able to modulate impulsivity in obese participants.

DETAILED DESCRIPTION:
In this single-blind, sham controlled study, the investigators will assess whether transcranial direct current stimulation (tDCS; a safe non-invasive method for modulating the activity of specific brain regions) when applied over the orbitofrontal cortex (OFC) is able to modulate impulsivity in obese volunteers. The investigators hypothesize that tDCS applied to the OFC, in comparison to sham tDCS, will significantly reduce impulsivity and enhance decision making as measured by computerized neurocognitive tasks. For this study the investigators will enroll 30 obese individuals aged 18-65 years. Participants will be assessed with a battery of computerized tasks as well as self-reported questionnaires on eating, impulsivity, mood and anxiety. Assessments will be carried out before, during, and after a single 20-minute 2mA tDCS session.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women aged 18 to 65
* have body mass index of 35 or above
* have had no recent change in medications in the 2 weeks prior participating in the study
* able to fast for 4 hours prior participating in the study

Exclusion Criteria:

* Active Substance use disorder
* Active Suicidal ideation
* Psychoactive Medication
* Past or current Gambling disorder
* Past or current Anorexia
* Past or current Bulimia Nervosa
* Past or current Psychosis
* Visual impairments preventing performance of the neuropsychological tasks
* Epilepsy
* Traumatic Brain Injury
* Stroke
* Neurological disorder affecting motor functions (Parkinsons, Huntington's, etc)
* Previous participation in tDCS research/treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Probabilistic Decision Making | Before and after a 20-minute tDCS session
  Net score of the Iowa Gambling Task The net score ranges from -20 to 30. Higher values represent a better outcome (i.e., enhanced decision-making)

SECONDARY OUTCOMES:
Cognitive Control | Before and after a 20-minute tDCS session
  Interference index in the Stroop Color-word Task. Interference index is the reaction time computed between the presentation of the stimulus and the response of the participant. It typically ranges from 0 to 300 millisecond, with smaller values of reaction time indicate better outcome (i.e., better cognitive control).
Food-specific cognitive control | Before and after a 20-minute tDCS session
  The interference index in the Food-Stroop Color-Word test. Interference index is the reaction time computed between the presentation of the stimulus and the response of the participant. It typically ranges from 0 to 300 millisecond, with smaller values of reaction time indicate better outcome (i.e., better Food-specific cognitive control).
Delayed discounting | Before and after a 20-minute tDCS session
  The discount rate for delayed monetary rewards. This rate is quantified by the hyperbolic discounting function using the following equation: V = A/(1+kD), where A presents the value of the delayed reward A at delay D, and k is a free parameter that determines the discount rate, with higher values of k indicate worse outcome (i.e., greater discounting of rewards as a function of time).
Motor impulsivity | Before and after a 20-minute tDCS session.
  The stop-signal reaction time in the Stop-Signal Task. The stop signal reaction time ranges from 50 to 250, where greater values represent worse outcome (i.e, increased motor impulsivity).
Moderation of effect by self-reported measures of impulsivity and dysregulated eating | Before and after a 20-minute tDCS session.
  Individuals with high levels of impulsivity, impulsive eating, binge eating, self-reported food addiction will show greater moderation by tDCS on our primary and secondary outcomes. Barrat's impulsiveness scale-11 with a range of scores from 0 to 120, with higher scores indicating greater impulsivity. Reward-based eating drive scale-13 with a range of scores from 0 to 54, with higher scores indicating greater uncontrolled eating. Binge eating scale with a range of scores from 0 to 46: minimal binge eating ( >17), moderate binge eating (18-26), and severe binge eating (<27)). Yale Food Addiction Scale with a range of symptom severity from 0 to 7: mild (2-3 symptoms), moderate (4-5 symptoms), severe (6 or more symptoms)).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Kringelbach ML. The human orbitofrontal cortex: linking reward to hedonic experience. Nat Rev Neurosci. 2005 Sep;6(9):691-702. doi: 10.1038/nrn1747. PMID 16136173
- [Background] Mason AE, Vainik U, Acree M, Tomiyama AJ, Dagher A, Epel ES, Hecht FM. Improving Assessment of the Spectrum of Reward-Related Eating: The RED-13. Front Psychol. 2017 May 30;8:795. doi: 10.3389/fpsyg.2017.00795. eCollection 2017. PMID 28611698
- [Background] Finlayson G, King N, Blundell J. The role of implicit wanting in relation to explicit liking and wanting for food: implications for appetite control. Appetite. 2008 Jan;50(1):120-7. doi: 10.1016/j.appet.2007.06.007. Epub 2007 Jun 28. PMID 17655972
- [Background] Nijs IM, Franken IH, Muris P. The modified Trait and State Food-Cravings Questionnaires: development and validation of a general index of food craving. Appetite. 2007 Jul;49(1):38-46. doi: 10.1016/j.appet.2006.11.001. Epub 2006 Dec 21. PMID 17187897
- [Background] O'Doherty JP, Deichmann R, Critchley HD, Dolan RJ. Neural responses during anticipation of a primary taste reward. Neuron. 2002 Feb 28;33(5):815-26. doi: 10.1016/s0896-6273(02)00603-7. PMID 11879657
- [Background] Ouellet J, McGirr A, Van den Eynde F, Jollant F, Lepage M, Berlim MT. Enhancing decision-making and cognitive impulse control with transcranial direct current stimulation (tDCS) applied over the orbitofrontal cortex (OFC): A randomized and sham-controlled exploratory study. J Psychiatr Res. 2015 Oct;69:27-34. doi: 10.1016/j.jpsychires.2015.07.018. Epub 2015 Jul 17. PMID 26343591
- [Background] Phelan S, Hassenstab J, McCaffery JM, Sweet L, Raynor HA, Cohen RA, Wing RR. Cognitive interference from food cues in weight loss maintainers, normal weight, and obese individuals. Obesity (Silver Spring). 2011 Jan;19(1):69-73. doi: 10.1038/oby.2010.138. Epub 2010 Jun 10. PMID 20539296
- [Background] Pursey KM, Stanwell P, Callister RJ, Brain K, Collins CE, Burrows TL. Neural responses to visual food cues according to weight status: a systematic review of functional magnetic resonance imaging studies. Front Nutr. 2014 Jul 9;1:7. doi: 10.3389/fnut.2014.00007. eCollection 2014. PMID 25988110
- [Background] Ray MK, Sylvester MD, Osborn L, Helms J, Turan B, Burgess EE, Boggiano MM. The critical role of cognitive-based trait differences in transcranial direct current stimulation (tDCS) suppression of food craving and eating in frank obesity. Appetite. 2017 Sep 1;116:568-574. doi: 10.1016/j.appet.2017.05.046. Epub 2017 May 29. PMID 28572072
- [Background] Rothemund Y, Preuschhof C, Bohner G, Bauknecht HC, Klingebiel R, Flor H, Klapp BF. Differential activation of the dorsal striatum by high-calorie visual food stimuli in obese individuals. Neuroimage. 2007 Aug 15;37(2):410-21. doi: 10.1016/j.neuroimage.2007.05.008. Epub 2007 May 18. PMID 17566768
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Swinburn B, Sacks G, Ravussin E. Increased food energy supply is more than sufficient to explain the US epidemic of obesity. Am J Clin Nutr. 2009 Dec;90(6):1453-6. doi: 10.3945/ajcn.2009.28595. Epub 2009 Oct 14. PMID 19828708
- [Background] van der Laan LN, de Ridder DT, Viergever MA, Smeets PA. The first taste is always with the eyes: a meta-analysis on the neural correlates of processing visual food cues. Neuroimage. 2011 Mar 1;55(1):296-303. doi: 10.1016/j.neuroimage.2010.11.055. Epub 2010 Nov 25. PMID 21111829